CLINICAL TRIAL: NCT03559205
Title: Implementing the MSK-HQ to Empower Patients and Improve Services
Brief Title: The MSK-Tracker Study
Acronym: MSK-Tracker
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keele University (Other)
Collaborators: Pro-Mapp Limited Company number 10152526 (Industry); Georgina Craig Associates Limited (Other); University of Oxford (Other); Arthritis Research UK (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: RG-0132-16-IPCHS
Record Dates: First submitted 2018-04-17; First posted 2018-06-18 (Actual); Results first posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-10

CONDITIONS: Musculoskeletal Pain
Keywords: Musculoskeletal; MSK
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Intervention Model Description: Before and after comparative study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MSK-Tracker (before) (No Intervention): Before - (Usual care in clinic consultations)
- MSK-Tracker (after) (Active Comparator): After - (MSK-Tracker in clinic consultations)
  Interventions: Other: MSK-Tracker

INTERVENTIONS:
Other: MSK-Tracker — The intervention is not a treatment, but involves patients and clinicians engaging with the MSK-Tracker software which will facilitate a new care planning approach with the following distinct components:
  * Pre-clinic preparation.
  * Clinic dashboard.
  * Summary action plan.
  * Personal goal setting.
  * Follow-up and monitoring.
  Arms: MSK-Tracker (after)

SUMMARY:
This study will co-design and test the feasibility and impact of implementing the Arthritis Research UK Musculoskeletal Health Questionnaire (MSK-HQ) using an e-PROM (electronic Patient Reported Outcome Measure) delivered via a digital health platform, with innovative embedded components called the MSK-Tracker. The MSK-Tracker uses the MSK-HQ as a foundation to help patients with MSK pain to:

* track the extent to which they are affected by their MSK condition across different aspects of their health,
* prepare appropriately for their clinical encounters, and
* take the right steps to making positive changes to improve their quality of life and manage their condition over the longer-term.

The Study Aims to:

1. Test the ability of the MSK-Tracker to act as an empowerment tool and method of facilitating a person-centred care planning approach in routine MSK clinic consultations.
2. Assess the value of the MSK-Tracker in generating aggregated outputs that inform MSK service improvement.

Study Design This study will use a before and after single Centre design with the comparator between phases 1 and 3 across a range of outcomes. Phase 2 will focus on iterative testing of the MSK-Tracker.

In addition, in Phase 1 and 3 will include qualitative research (site 1 only) using the Experience Based Co-Design (EBCD) methodology to explore the impact of the MSK-Tracker and to inform further improvement and refinement of the tool and its use within the context of an MSK service and clinical practice. The findings from the qualitative research will be triangulated with insights from the aggregated data of patient outcomes to enrich and help make sense of the study findings.

DETAILED DESCRIPTION:
The Arthritis Research UK Musculoskeletal Health Questionnaire (MSK-HQ) is a recently validated new MSK Patient Reported Outcome Measure (PROM) that has been co-produced with patients and clinicians to measure the holistic impact of an MSK condition on a person's health. It has been validated in both primary and secondary care populations and is appropriate for use by patients across the care pathway. It is designed for use in routine, busy, clinical practice. The MSK-HQ is freely available to the NHS, and consists of 14 health items that cover the domains that matter the most to MSK patients and helps clinicians and patients to identify the areas of life where the condition is impacting most. An electronic-PROM (e-PROM) version of the MSK-HQ is available and is being used by some early adopter MSK services to audit their clinical and patient outcome performance.

However, it is not yet known whether:

* Patients using the MSK-HQ routinely as part of their care planning, supports them to feel more involved and empowered in managing their health issues.
* Using the MSK-HQ can facilitate a more holistic care planning consultation, both in terms of the quality of patient interactions and communications with healthcare professionals.
* It is acceptable or feasible for both patients and clinicians to use the MSK-HQ as an e-PROM.

Enabling organisations to examine their aggregated MSK-HQ data at service level identifies unmet need, improvement opportunities and informs MSK service and organisational developments.

This research will optimise implementation of the MSK-HQ using a digital health platform, and evaluate its impact on both clinicians and patients. In addition to investigating benefits at the individual level, we also hypothesise that the data generated by this innovation may provide substantial organisational level insight. We plan therefore to explore how MSK-HQ data can best be aggregated, made sense of and presented as actionable outputs that identify unmet need and service improvement opportunities.

This proposal is novel because of three specific developments;

i. The development of an IT innovation to support the implementation of the MSK-HQ within the individual consultation, which has the potential to bring many advantages to people with MSK conditions. The individual patient is often the only consistent connection between different service components. It therefore makes sense for patients to be able to own and access their care plan as they move between providers. For conditions such as osteoarthritis, many core treatments are initiated by patients themselves rather than by the doctor and the perspectives of patients may differ from the perspectives of healthcare professionals, with information recorded by professionals in the medical records not necessarily aligned to the patient's ideas about his or her treatment plan.

ii. Making the MSK-HQ available to patients in advance as a prompt prior to their consultations, and testing if its application in this way facilitates a care planning approach. Patients want to be able to own and access their care plan as they move between providers, and the MSK-Tracker will enable them to do that. Patients can also find it difficult to raise important issues of concern in short, busy clinical interactions with different providers, which can lead to healthcare inconsistencies and inequalities in the support they receive. Although reports are limited, evidence from cancer research suggests that the use of consultation prompt lists can improve care and augment consultations when they are used proactively by clinicians. Despite growing evidence that they can make the consultation more focused and time-efficient, prompt lists are infrequently used in NHS MSK consultations. Within the UK health community, there is a national debate about how to bring about more person-centred care "How can we get better at providing patient centred care?", and "No decision about me without me". Participants in the BMJ discussion agreed that a change in culture and better use of technology could benefit patients and doctors. The potential for the MSK-Tracker to influence the consultation and help patients keep track of their health status and in control of their care resonates with the 2014 Reith Lectures by Atul Gawande, who highlighted the role of checklists and prompt questions as a stimulus for achieving better outcomes and service improvement. Problems with 'the system': the interactions between people and organisations that deliver healthcare were also highlighted. This debate is of growing relevance to the MSK community and new national policy from Arthritis Research UK is now focused on efforts to ensure that those living with arthritis and musculoskeletal conditions get the care and support they need to lead as healthy and active a life as possible in order to be "In control, independent and recognised". It is clear that to empower patients to feel well supported, informed and able to manage the effects of their condition and minimise its impact on their lives, they need to have equal voice and be at the heart of setting goals and planning their own care in partnership with their MSK clinical team. However, in order to deliver changes to the way care is delivered, innovative technological solutions such as this, are required.

iii. Identifying the best ways to present and format outputs of aggregated MSK-HQ data to generate insights that inform service development and improvement. The MSK-Tracker will be an exciting new development, which, if implemented through a scalable electronic solution, has substantial potential to drive forward large scale service changes. MSK-HQ is supported nationally by Arthritis Research UK, NHS England and professional bodies including the CSP (Chartered Society of Physiotherapy) and BOA (British Orthopaedic Association). The next important step is to find a feasible way to use this outcome measure within routine clinical practice as a stimulus to drive the whole system to focus on what matters to patients and improve the care provided.

The study is using a 'before' and 'after' sequential comparison design with an iterative pilot and user testing phase in between. In addition, audio recordings of the consultation (site 1 only) (in a sub-sample, n=40 (phase 1=20 & phase 3=20)), alongside individual clinician and patient interviews and a feedback workshop with clinicians and patients, will explore the feasibility, and impact of implementing the MSK-Tracker within routine consultations and the experiences of those who have used it.

Phase 1 ('Before' stage). Patients (n=200) who meet the eligibility criteria for having long-term MSK pain and an appointment at the relevant clinic will be consented and recruited to complete the e-PROM survey and demographic information shortly before their consultation. This phase will seek to collect patient information via the online digital health platform without using the new innovative 'MSK-Tracker' components, in order to give a baseline of what changes are observed before the MSK-Tracker intervention is used. Patients will complete data online before clinic, and then 2 weeks and 3 months after clinic and their change scores examined. Clinicians will complete a case report form (CRF) using the clinician portal to record clinical behaviours within the consultation. Audio recordings of approximately 20 patient consultations will examine consultation conversations and their content (site 1 only).

Phase 2. ('Pilot stage') (Site 1 only). The MSK-Tracker will be developed and optimised through an iterative user testing framework with patients, clinicians, software provider, and experts. The MSK-Tracker will have a number of key 'care planning' components including, pre-clinic preparation, clinic dashboard, summary action plan, personal goal setting and follow-up and progress charts.

Early pilot testing of the MSK-Tracker will mirror the processes used in phase 3, with a limited number of patients and clinicians using the Tracker. The aim is to recruit approximately 40 patients (in 2 cycles of 20) to use the MSK-Tracker. During this phase all patients and clinicians will be invited to take part in an interview about their experiences to identify further potential improvements that can be made to the Tracker before commencing phase 3. The aim is to interview up to 10 patients in each of the 2 cycles.

Phase 3 ('After' stage). Identical to phase 1, patients (n=200) who meet the eligibility criteria for having long-term MSK pain and an appointment at a relevant clinic, will complete an e-PROM shortly before their consultation and again 2 weeks and 3 months after their consultation. During phase 3 the MSK-Tracker components will be used alongside the e-PROM to support the new innovative 'care planning' approach and clinicians will be trained to use the MSK-Tracker within their clinical encounters. As in phase 1 audio recordings of approximately 20 patient consultations (site 1 only) will examine consultation conversations and their content. A descriptive content analysis will be conducted to identify differences before and after the introduction of the MSK-Tracker in clinic.

In addition, qualitative research will take place using the Experience Based Co-Design (EBCD) methodology in both phase 1 and 3 (site 1 only). This will involve interviews with approximately 10 patients and up to 10 clinicians to explore the impact of the MSK-Tracker and to inform further improvement and refinement of the tool and its use within the context of an MSK service and clinical practice. The findings from this qualitative research will be triangulated with insights from the aggregated data of patient outcomes to enrich and help make sense of the study findings.

The intervention is not a treatment per se, but involves patients and clinicians engaging with the MSK-Tracker software. It is envisaged that the MSK-Tracker will facilitate a new care planning approach with the following distinct components:

* Pre-clinic preparation. Prior to a consultation, the MSK-Tracker will help patients to set their clinic agenda by asking them to think about the ways in which their long-term MSK condition is impacting on their lives.
* Clinic dashboard. During the consultation it will enable the clinician to see the patient's health impact from their MSK condition (using MSK-HQ), and present the patient's clinic agenda to inform the consultation focus and ensure the individual's specific needs are addressed.
* Summary action plan. The Tracker will be used to record the agreed action plan from the consultation, including advice, information, referrals and investigations, which the patient can access when they want to as a reminder of what was agreed.
* Personal goal setting. To help the patient focus on what they personally seek to change (e.g. to get more fit and active) in relation to the impact of the MSK condition on their life and to help them reflect on what things are helping/hindering them to achieve goals to reduce this impact a goal setting module will be available to patients within the Tracker.
* Follow-up and monitoring. The Tracker will enable the patient to re-take the MSK-HQ at 2 weeks and 3 months and then have the opportunity to look at tracker charts that show their progress on the MSK-HQ overall score and individual domains.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and above with an appointment to attend the Staffordshire Musculoskeletal Interface Service for an MSK pain problem will be invited to take part.

Exclusion Criteria:

* Patients unable to use or access the internet will be unable to take part in this research as well as patients who do not provide informed consent for study participation and data collection. The online system will only be available in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Hill, Dr, Principal Investigator — Keele University
Locations (1):
- Haywood Hospital, Stoke-on-Trent, Staffordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Note 321 participants were enrolled but baseline data was only collected from 273.
Groups:
- MSK-Tracker (Before): Usual Care in clinic consultations
- MSK-Tracker (After): Use of the MSK-Tracker in clinic consultations
  MSK-Tracker: The intervention is not a treatment, but involves patients and clinicians engaging with the MSK-Tracker software which will facilitate a new care planning approach with the following distinct components:
  * Pre-clinic preparation.
  * Clinic dashboard.
  * Summary action plan.
  * Personal goal setting.
  * Follow-up and monitoring.
Period: Overall Study
Arm/Group | MSK-Tracker (Before) | MSK-Tracker (After)
Started | 177 | 144
Baseline Data | 141 | 132
Completed | 65 | 57
Not Completed | 112 | 87

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MSK-Tracker (Before) | MSK-Tracker (After) | Total
Number analyzed (Participants) | 141 | 132 | 273
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.73 (15.06) | 51.91 (14.61) | 53.88 (14.94)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 74 | 81 | 155
  Female | 67 | 50 | 117
  Prefer not to say | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Mixed | 1 | 1 | 2
  Asian | 3 | 2 | 5
  Black | 2 | 0 | 2
  White | 133 | 126 | 259
  Other | 1 | 2 | 3
  Prefer not to say | 1 | 1 | 2
  Missing | 0 | 0 | 0
Pain Location(s) [Number; unit: Participants]
  Head region | 3 | 3 | 6
  Neck | 27 | 27 | 54
  Shoulder/upper arm | 35 | 27 | 62
  Lower arm/wrist | 16 | 11 | 27
  Hand(s) | 14 | 19 | 33
  Upper back/chest/abdomen | 13 | 14 | 27
  Lower back/pelvis | 64 | 59 | 123
  Hip, groin, thigh | 39 | 36 | 75
  Knee/lower leg | 42 | 51 | 93
  Ankle/foot | 22 | 28 | 50
  Other | 12 | 9 | 21
Problem duration [Count of Participants; unit: Participants]
  < 2 weeks | 0 | 0 | 0
  2 to 4 weeks | 6 | 2 | 8
  5 weeks to 3 months | 32 | 18 | 50
  4 to 6 months | 21 | 14 | 35
  7 to 12 months | 16 | 21 | 37
  13 months to 3 years | 35 | 30 | 65
  > 3 years | 30 | 46 | 76
  Missing | 1 | 1 | 2
Previous physio for problem [Count of Participants; unit: Participants]
  No | 65 | 77 | 142
  Yes | 76 | 55 | 131
Previous surgery for problem [Count of Participants; unit: Participants]
  No related surgery | 124 | 116 | 240
  1 related surgery | 11 | 8 | 19
  2 related surgeries | 3 | 4 | 7
  3 or more related surgeries | 3 | 4 | 7
  Missing | 0 | 0 | 0
Referral source [Count of Participants; unit: Participants]
  GP | 130 | 126 | 256
  Self-referral | 0 | 1 | 1
  Orthopaedic Surgeon | 7 | 1 | 8
  Neurologist/Neurosurgeon | 1 | 0 | 1
  Occupational Health | 3 | 4 | 7
  Other | 0 | 0 | 0
  Missing | 0 | 0 | 0
Comorbidities: [Number; unit: participants]
  Heart disease | 45 | 4 | 49
  High blood pressure | 39 | 34 | 73
  Poor circulation | 19 | 16 | 35
  Lung disease | 3 | 7 | 10
  Diabetes | 15 | 13 | 28
  Kidney disease | 1 | 2 | 3
  Neurological disorder | 1 | 7 | 8
  Liver disease | 0 | 1 | 1
  Cancer | 3 | 4 | 7
  Depression | 29 | 37 | 66
  Arthritis | 41 | 36 | 77
  None | 55 | 46 | 101
Number of Comorbidities [Mean (Standard Deviation); unit: Comorbidities] | 1.55 (1.01) | 1.57 (1.01) | 1.56 (1.01)
Independence [Number; unit: participants]
  Needed assistance to fill in this questionnaire | 8 | 13 | 21
  Considers self to have a carer | 11 | 19 | 30
Health Literacy - Help needed to read instructions [Number; unit: participants] | 5 | 8 | 13
Work status - Working [Number; unit: Participants] | 75 | 73 | 148
Hours missed from work in last 7 days because of problem [Mean (Standard Deviation); unit: Hours] — Population: only working patients
  Hours
    number analyzed (Participants) | 75 | 73 | 148
    (all) | 9.13 (21.24) | 8.49 (31.67) | 8.81 (26.8)
Hours missed from work in last 7 days for other reasons [Mean (Standard Deviation); unit: Hours] — Population: only working patients
  Hours
    number analyzed (Participants) | 75 | 73 | 148
    (all) | 8.05 (33.46) | 11.45 (36.82) | 9.73 (35.08)
Hours worked in last 7 days [Mean (Standard Deviation); unit: Hours] — Population: only working patients
  Hours
    number analyzed (Participants) | 75 | 73 | 148
    (all) | 28.11 (18.74) | 25.29 (15.21) | 26.72 (17.09)
Joint and muscle symptoms affect productivity [Mean (Standard Deviation); unit: units on a scale] — The response to the question "During the past seven days, how much did your joint and muscle symptoms affect your productivity while you were working?"
  0-10 integer scale where:
  0 = Joint and muscle symptoms had no effect on my work 10 = Joint and muscle symptoms completely prevented me from working Population: only working patients
  units on a scale
    number analyzed (Participants) | 75 | 73 | 148
    (all) | 4.81 (2.26) | 5.21 (1.88) | 5.02 (2.07)
Joint and muscle symptoms affect ability to do regular daily activities, other than work [Mean (Standard Deviation); unit: units on a scale] — The response to the question "During the past seven days, how much did your joint and muscle symptoms affect your ability to do your regular daily activities, other than work at a job?"
  0-10 integer scale where:
  0 = Joint and muscle symptoms had no effect on my daily activities 10 = Joint and muscle symptoms completely prevented me from doing my daily activities Population: only working patients
  units on a scale
    number analyzed (Participants) | 75 | 73 | 148
    (all) | 5.61 (2.19) | 5.71 (2.03) | 5.66 (2.10)
Percent work time missed due to problem [Mean (Standard Deviation); unit: Percentage of work time] — Population: Working only excluding missing
  Percentage of work time
    number analyzed (Participants) | 66 | 68 | 134
    (all) | 22 (36) | 16 (30) | 19 (33)
Percent impairment while working due to problem [Mean (Standard Deviation); unit: Percentage of impairment] — Population: Working only excluding missing
  Percentage of impairment
    number analyzed (Participants) | 58 | 63 | 121
    (all) | 48 (23) | 52 (16) | 50 (21)
Percent overall work impairment due to problem [Mean (Standard Deviation); unit: percentage of overall work impairment] — Population: Working only excluding missing
  percentage of overall work impairment
    number analyzed (Participants) | 57 | 63 | 120
    (all) | 52 (25) | 56 (20) | 54 (22)
Percent activity impairment due to problem [Mean (Standard Deviation); unit: percentage of activity impairment] — Population: Working only excluding missing
  percentage of activity impairment
    number analyzed (Participants) | 75 | 73 | 148
    (all) | 56 (22) | 57 (20) | 57 (21)

OUTCOME MEASURES:

1. Primary Outcome: Patient Enablement Instrument (PEI)
Description: A measure of patient empowerment.
  Scale:
  Much better / Much more = 2 Better / More = 1 Same or less = 0 Not applicable = 9
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MSK-Tracker (Before) | MSK-Tracker (After)
Number analyzed (Participants) | 75 | 66
units on a scale | 1.48 (1.97) | 1.50 (2.31)
Statistical Analysis 1: Comparison: MSK-Tracker (Before) vs MSK-Tracker (After); 2 Week Analysis; Test type: Superiority; p = 0.96, t-test, 2 sided; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.74 to 0.70]

2. Secondary Outcome: Musculoskeletal Health Questionnaire (MSK-HQ)
Description: This questionnaire is about joint, back, neck, bone and muscle symptoms such as aches, pains and/or stiffness.
  Min score = 0; Max score = 56. A higher score indicates better outcome.
Time Frame: Baseline, 2 weeks and 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MSK-Tracker (Before) | MSK-Tracker (After)
Number analyzed (Participants) | 141 | 132
units on a scale
  Baseline | 24.32 (8.26) | 24.45 (9.83)
  2-week | 26.63 (9.50) | 24.62 (10.09)
  3-month | 27.17 (10.61) | 26.23 (11.02)
Statistical Analysis 1: Comparison: MSK-Tracker (Before) vs MSK-Tracker (After); Baseline; Test type: Superiority; p = 0.90, t-test, 2 sided; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-2.31 to 2.04]
Statistical Analysis 2: Comparison: MSK-Tracker (Before) vs MSK-Tracker (After); 2 Week Analysis; Test type: Superiority; p = 0.21, t-test, 2 sided; Mean Difference (Final Values) = 2.01, 95% CI 2-sided [-1.17 to 5.19]
Statistical Analysis 3: Comparison: MSK-Tracker (Before) vs MSK-Tracker (After); 3-Month; Test type: Superiority; p = 0.63, t-test, 2 sided; Mean Difference (Final Values) = 0.94, 95% CI 2-sided [-2.95 to 4.83]

3. Secondary Outcome: Consumer Health Activation Index (CHAI)
Description: The CHAIv1 was developed for use among diverse patients to provide a measure of patient activation.
  Min score = 0, Max score = 100. A high score represents a better outcome.
  "low" (CHAI score 0-79), "moderate" (CHAI score 80-94), and "high" (CHAI score 95-100).
Time Frame: Baseline, 2 weeks and 3 months
Population: Loss to follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MSK-Tracker (Before) | MSK-Tracker (After)
Number analyzed (Participants) | 141 | 132
units on a scale
  Baseline | 71.42 (15.8) | 68.79 (14.68)
  2-weeks: number analyzed (Participants) | 82 | 70
  2-weeks | 73.24 (12.65) | 71.03 (13.61)
  3-months: number analyzed (Participants) | 64 | 57
  3-months | 72.72 (15.02) | 72.14 (12.25)
Statistical Analysis 1: Comparison: MSK-Tracker (Before) vs MSK-Tracker (After); Baseline; Test type: Superiority; p = 0.15, t-test, 2 sided; Mean Difference (Final Values) = 2.63, 95% CI 2-sided [-1.00 to 6.26]
Statistical Analysis 2: Comparison: MSK-Tracker (Before) vs MSK-Tracker (After); Week 2 analysis; Test type: Superiority; p = 0.30, t-test, 2 sided; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [-2.02 to 6.45]
Statistical Analysis 3: Comparison: MSK-Tracker (Before) vs MSK-Tracker (After); 3-Month; Test type: Superiority; p = 0.85, t-test, 2 sided; Mean Difference (Final Values) = 0.50, 95% CI 2-sided [-4.89 to 5.90]

4. Secondary Outcome: Valuing Patients as Individuals Scale (Short Version)
Description: Scale 1 - Care and Respect Min score = 0, Max score = 15 Higher score indicates a better outcomes.
  Scale 2 - Understanding and Engagement:
  Min score = 0, Max score = 15. Higher score indicates a better outcomes.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MSK-Tracker (Before) | MSK-Tracker (After)
Number analyzed (Participants) | 80 | 70
units on a scale
  Care and respect | 13.1 (2.13) | 12.99 (1.75)
  Understanding & engagement | 12.71 (2.18) | 12.49 (1.55)
Statistical Analysis 1: Comparison: MSK-Tracker (Before) vs MSK-Tracker (After); Care and respect; Test type: Superiority; p = 0.72, t-test, 2 sided; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.51 to 0.74]
Statistical Analysis 2: Comparison: MSK-Tracker (Before) vs MSK-Tracker (After); Understanding & engagement; Test type: Superiority; p = 0.46, t-test, 2 sided; Mean Difference (Final Values) = 0.23, 95% CI 2-sided [-0.38 to 0.83]

5. Secondary Outcome: Global Rating of Change (1 Item)
Description: The response to the question:
  "With respect to your joint and muscle symptoms, how would you describe yourself now compared to how it was when you came to the Haywood clinic?"
  Much better = 5 Better = 4 Same = 3 Worse = 2 Much worse = 1 Prefer not to say = 9
Time Frame: 2 weeks and 3 months
Population: Loss to follow up
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | MSK-Tracker (Before) | MSK-Tracker (After)
Number analyzed (Participants) | 82 | 70
Score
  2-weeks | 2.91 (0.74) | 2.71 (0.68)
  3-months: number analyzed (Participants) | 63 | 57
  3-months | 2.98 (1.01) | 2.82 (0.97)
Statistical Analysis 1: Comparison: MSK-Tracker (Before) vs MSK-Tracker (After); 2-weeks; Test type: Superiority; p = 0.30, t-test, 2 sided; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [-0.13 to 0.42]
Statistical Analysis 2: Comparison: MSK-Tracker (Before) vs MSK-Tracker (After); 3-months; Test type: Superiority; p = 0.38, t-test, 2 sided; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [-0.20 to 0.52]

6. Secondary Outcome: The Patient Enablement Scale
Description: A measure of patient empowerment
  Min score = 0, Max score = 12. Higher score indicated better outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MSK-Tracker (Before) | MSK-Tracker (After)
Number analyzed (Participants) | 62 | 56
units on a scale | 1.82 (2.12) | 2.12 (3.33)
Statistical Analysis 1: Comparison: MSK-Tracker (Before) vs MSK-Tracker (After); Test type: Superiority; p = 0.61, t-test, 2 sided; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-1.48 to 0.88]

ADVERSE EVENTS:
Time Frame: Up to 1 year from baseline data collection.
Description: Note that only participants who provided baseline data were monitored for adverse events.
Arm/Group | MSK-Tracker (Before) | MSK-Tracker (After)
All-Cause Mortality (participants affected / at risk) | 0/141 | 0/132
Serious Adverse Events (participants affected / at risk) | 0/141 | 0/132
Other Adverse Events (participants affected / at risk) | 0/141 | 0/132

LIMITATIONS AND CAVEATS:
This project was limited to a single clinical site and to the specific context of an interface clinic setting in between community care and secondary care services within the NHS.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-12-10): https://cdn.clinicaltrials.gov/large-docs/05/NCT03559205/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/05/NCT03559205/SAP_001.pdf